CLINICAL TRIAL: NCT01586364
Title: Long-Term Safety of Ospemifene 60 mg Oral Daily Dose for the Treatment of Vulvar and Vaginal Atrophy (VVA) in Postmenopausal Women Without a Uterus: A 52-Week Open-Label Follow-Up to Protocol 15-50310
Brief Title: Long-Term Safety of Ospemifene 60 mg Oral Daily Dose for the Treatment of Vulvar and Vaginal Atrophy (VVA) in Postmenopausal Women Without a Uterus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Collaborators: QuatRx Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-50312
Record Dates: First submitted 2012-04-18; First posted 2012-04-26 (Estimated); Results first posted 2013-06-28 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-04

CONDITIONS: Atrophy; Vaginal Diseases
Keywords: Menopausal symptoms; Vulvar and vaginal atrophy in menopausal women; Vaginal atrophy; Urogenital atrophy
MeSH Terms: conditions — Atrophy; Vaginal Diseases | interventions — Ospemifene; Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ospemifene 60 mg Oral Tablet (Experimental): Participants will take one tablet of ospemifene 60 mg orally, once a day for 12 weeks.
  Interventions: Drug: Ospemifene 60Mg Oral Tablet

INTERVENTIONS:
Drug: Ospemifene 60Mg Oral Tablet
  Other Names: Osphena®

SUMMARY:
The objective of the study was to assess the long-term safety of daily doses of ospemifene 60 mg in the treatment of vulvar and vaginal atrophy (VVA) in postmenopausal women without a uterus.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 40 to 80 years with a diagnosis of vulvar and vaginal atrophy (VVA) as assessed by vaginal pH, maturation index of vaginal smear, and self-reported symptoms at Baseline for Protocol 15-50310
* Did not have a uterus
* Met the inclusion and exclusion criteria for Protocol 15-50310
* Had completed Protocol 15-50310 without any clinically significant abnormal findings at the end-of-study visit for Protocol 15-50310
* Provided written informed consent to participate in the study and agreed to follow dosing instructions and complete all required study visits

Exclusion Criteria:

* Had clinically significant abnormal findings at the Week 12 End of Study visit for Protocol 15-50310
* Had any physical or mental condition which, in the opinion of the investigator, may have interfered with the subject's ability to comply with the study procedures

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2006-05-08 (Actual); Primary Completion 2008-11-21 (Actual); Study Completion 2008-12-22 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm = 60 mg Ospemifene: Subjects took an oral dose of Ospemifene 60 mg tablet each morning with food for 52 weeks
Period: Overall Study
Arm/Group | Treatment Arm = 60 mg Ospemifene
Started | 301
Completed | 184
Not Completed | 117
Not completed — Withdrawal by Subject | 40
Not completed — Adverse Event | 37
Not completed — Lost to Follow-up | 17
Not completed — Protocol Violation | 16
Not completed — Lack of Efficacy | 1
Not completed — Other-Did not feel better post-treatment | 1
Not completed — Other-Subject wasn't getting much relief | 1
Not completed — Other-Site closure due to PI illness | 1
Not completed — Other-PI discretion, site closing | 2
Not completed — Other-Not specified | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 301
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (6.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 301
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 280
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 278
  Black or African American | 11
  Asian | 6
  American Indian or Alaska Native | 3
  Other | 3
Height [Mean (Standard Deviation); unit: cm] | 161.90 (6.026)
Weight [Mean (Standard Deviation); unit: kg] | 70.54 (13.024)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.865 (4.4106)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs)
Time Frame: Week 13 (Phone Contact) to Week 56 (Visit 4)
Measure: Number; unit: Participants
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 301
Participants
  Treatment-Emergent AE | 220
  Related AE (Possibly/Probably/Definitely Related) | 67
  AE Causing Study Drug Discontinuation | 34
  Serious AE | 13
  Severe AE | 38

2. Primary Outcome: Change From Baseline in Serum Lipid Levels at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: The ITT population was used for the analysis. For this particular outcome measure, 241 out of 301 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 241
percent change
  Total Cholesterol | 1.59 (17.772)
  Low-density lipoprotein cholesterol (LDL-C) | 2.83 (29.420)
  High-density lipoprotein cholesterol (HDL-C) | 2.81 (16.009)
  Triglycerides | 11.51 (43.422)

3. Primary Outcome: Change From Baseline in Serum Lipid Levels at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: The ITT population was used for the analysis. For this particular outcome measure, 195 out of 301 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 195
percent change
  Total Cholesterol | -0.02 (16.025)
  LDL-C | -0.54 (22.932)
  HDL-C | 2.74 (15.226)
  Triglycerides | 13.07 (43.877)

4. Primary Outcome: Change From Baseline in Blood Pressure at Visit 2
Description: Systolic blood pressure (SBP), diastolic blood pressure (DBP)
Time Frame: Baseline to Week 26 (Visit 2)
Population: The ITT population was used for the analysis. For this particular outcome measure, at week 26, 244 out of 301 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 244
mmHg
  SBP | -1.2 (15.91)
  DBP | -0.7 (9.32)

5. Primary Outcome: Change From Baseline in Pulse Rate at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 244
bpm | 2.1 (10.22)

6. Primary Outcome: Change From Baseline in Weight at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 244
kg | 0.798 (3.6022)

7. Primary Outcome: Change From Baseline in Body Mass Index (BMI) at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 244
kg/m^2 | 0.309 (1.3628)

8. Primary Outcome: Change From Baseline in Blood Pressure at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: The ITT population was used for the analysis. For this particular outcome measure, at week 52, 199 out of 301 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 199
mmHg
  SBP | -1.2 (16.35)
  DBP | -1.0 (9.88)

9. Primary Outcome: Change From Baseline in Pulse Rate at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 199
bpm | 3.3 (9.43)

10. Primary Outcome: Change From Baseline in Weight at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 199
kg | 1.122 (8.2464)

11. Primary Outcome: Change From Baseline in BMI at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 199
kg/m^2 | 0.439 (3.2779)

12. Primary Outcome: Change From Baseline in Visual Evaluation of Vagina at Visit 2
Description: Each of the categories in the table was assessed on a 4-point scale (0=None, 1=Mild, 2=Moderate, 3=Severe)
Time Frame: Baseline to Week 26 (Visit 2)
Population: The ITT population was used for the analysis. For this particular outcome measure, at week 26, 243 out of 301 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 243
units on a scale
  Petechiae | -0.6 (0.86)
  Pallor | -1.0 (0.95)
  Friability | -0.8 (0.89)
  Vaginal Dryness in Mucosa | -1.4 (0.87)
  Vaginal Redness in Mucosa | -0.6 (0.92)

13. Primary Outcome: Change From Baseline in Visual Evaluation of Vagina at Visit 3
Description: Each of the categories in the table was assessed on a 4-point scale (0=None, 1=Mild, 2=Moderate, 3=Severe)
Time Frame: Baseline to Week 52 (Visit 3)
Population: The ITT population was used for the analysis. For this particular outcome measure, at week 52, 198 out of 301 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 198
units on a scale
  Petechiae | -0.6 (0.90)
  Pallor | -1.2 (0.95)
  Friability | -0.8 (0.91)
  Vaginal Dryness in Mucosa | -1.5 (0.88)
  Vaginal Redness in Mucosa | -0.8 (0.89)

14. Primary Outcome: Assessment of Cervical Pap Smear Samples (if Cervix is Intact)
Description: Cervical Pap smear samples are used to evaluate: atypical squamous cells of undetermined significance (ASC-US), squamous intraepithelial lesions (SILs), intraepithelial lesions or malignancy, and reactive endocervical cells and/or metaplastic cells.
Time Frame: Week 52 (Visit 3)
Population: The ITT population was used for the analysis. For this particular outcome measure, at week 52, 16 out of 301 subjects were analyzed.
Measure: Number; unit: Participants
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 16
Participants
  Atypical Squamous Cells-Undetermined Significance | 1
  Negative for Intraepithelial Lesion or Malignancy | 15

15. Primary Outcome: Assessment of Breast Palpation at Visit 2
Description: Breast palpation was used to assess breast abnormalities.
Time Frame: Week 26 (Visit 2)
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 243
Participants
  Normal | 243
  Abnormal | 0

16. Primary Outcome: Assessment of Breast Palpation at Visit 3
Description: Breast palpation was used to assess breast abnormalities.
Time Frame: Week 52 (Visit 3)
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 199
Participants
  Normal | 198
  Abnormal | 1

17. Primary Outcome: Change From Baseline in Coagulation Parameters (Antithrombin Antigen, Protein C Antigen, Protein S Antigen) at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: The ITT population was used for the analysis. For this particular outcome measure, at week 26, 242 out of 301 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 242
percent change
  Antithrombin Antigen, Plasma | 0.4 (10.70)
  Protein C Antigen, Plasma | -1.3 (21.62)
  Protein S Antigen, Free, Plasma | 9.6 (15.19)

18. Primary Outcome: Change From Baseline in Activated Partial Thromboplastin Time (Plasma) at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 242
s | -1.5 (14.36)

19. Primary Outcome: Change From Baseline in Fibrinogen (Plasma) Levels at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 242
mg/dL | -25.4 (80.30)

20. Primary Outcome: Change From Baseline in Coagulation Parameters (Antithrombin Antigen, Protein C Antigen, Protein S Antigen) at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: The ITT population was used for the analysis. For this particular outcome measure, at week 52, 194 out of 301 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 194
percent change
  Antithrombin Antigen, Plasma | 2.4 (10.80)
  Protein C Antigen, Plasma | 4.3 (22.57)
  Protein S Antigen, Free, Plasma | 12.9 (20.40)

21. Primary Outcome: Change From Baseline in Activated Partial Thromboplastin Time (Plasma) at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 194
s | -0.7 (17.24)

22. Primary Outcome: Change From Baseline in Fibrinogen (Plasma) Levels at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 194
mg/dL | -29.9 (77.19)

23. Primary Outcome: Change From Baseline in Leukocyte, Lymphocyte, Monocyte and Platelet Count Levels at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: The ITT population was used for the analysis. For this particular outcome measure, at week 26, 240 out of 301 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: (x10(9)/L)
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 240
(x10(9)/L)
  Leukocytes | -0.17 (1.201)
  Lymphocytes | -0.058 (0.4025)
  Monocytes | -0.012 (0.1557)
  Platelet Count | -6.2 (41.68)

24. Primary Outcome: Change From Baseline in Erythrocyte Levels at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: (x10(12)/L)
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 240
(x10(12)/L) | -0.098 (0.2454)

25. Primary Outcome: Change From Baseline in Hemoglobin Levels at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 240
g/dL | -0.29 (0.705)

26. Primary Outcome: Change From Baseline in Hematocrit and Red Blood Cell (RBC) Distribution Width at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 240
percent change
  Hematocrit | -0.86 (2.151)
  RBC distribution width | 0.07 (0.776)

27. Primary Outcome: Change From Baseline in Mean Corpuscular Volume (MCV) and Mean Platelet Volume (MPV) at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 240
fL
  MCV, free | 0.02 (1.732)
  MPV | 0.01 (0.521)

28. Primary Outcome: Change From Baseline in Leukocyte, Lymphocyte, Monocyte and Platelet Count Levels at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: The ITT population was used for the analysis. For this particular outcome measure, at week 52, 196 out of 301 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: (x10(9)/L)
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 196
(x10(9)/L)
  Leukocytes | -0.05 (1.270)
  Lymphocytes | -0.010 (0.4410)
  Monocytes | -0.021 (0.1619)
  Platelet Count | -13.5 (36.92)

29. Primary Outcome: Change From Baseline in Erythrocyte Levels at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: (x10(12)/L)
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 196
(x10(12)/L) | -0.108 (0.2745)

30. Primary Outcome: Change From Baseline in Hemoglobin Levels at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 196
g/dL | -0.35 (0.840)

31. Primary Outcome: Change From Baseline in Hematocrit and RBC Distribution Width at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 196
percent change
  Hematocrit | -0.97 (2.490)
  RBC distribution width | 0.14 (0.834)

32. Primary Outcome: Change From Baseline in MCV and MPV at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 196
fL
  MCV, free | 0.01 (2.081)
  MPV | -0.03 (0.512)

33. Primary Outcome: Change From Baseline in Albumin and Total Protein Levels at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 243
g/dL
  Albumin, Serum | -0.10 (0.248)
  Total Protein, Serum | -0.14 (0.399)

34. Primary Outcome: Change From Baseline in Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Creatine Kinase (CK) Levels at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 243
U/L
  ALT, Serum | -3.7 (10.93)
  AST, Serum | -0.1 (5.62)
  CK, Serum | -6.7 (46.23)

35. Primary Outcome: Change From Baseline in Bilirubin, Creatinine, Glucose, Uric Acid and Blood Urea Nitrogen (BUN) Levels at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 243
mg/dL
  Bilirubin Total, Serum | -0.08 (0.144)
  Creatinine, Plasma/Serum | -0.06 (0.125)
  Glucose, Plasma/Serum | 3.2 (17.75)
  Uric Acid, Serum | -0.02 (0.786)
  BUN | 0.5 (3.86)

36. Primary Outcome: Change From Baseline in Albumin and Total Protein Levels at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: The ITT population was used for the analysis. For this particular outcome measure, at week 52, 197 out of 301 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 197
g/dL
  Albumin, Serum | -0.08 (0.232)
  Total Protein, Serum | -0.19 (0.376)

37. Primary Outcome: Change From Baseline in ALT, AST and CK Levels at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 197
U/L
  ALT, Serum | -4.1 (11.81)
  AST, Serum | 0.2 (7.06)
  CK, Serum | 2.6 (109.35)

38. Primary Outcome: Change From Baseline in Bilirubin, Creatinine, Glucose, Uric Acid and BUN Levels at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 197
mg/dL
  Bilirubin Total, Serum | -0.08 (0.151)
  Creatinine, Plasma/Serum | -0.04 (0.125)
  Glucose, Plasma/Serum | 3.6 (16.47)
  Uric Acid, Serum | 0.03 (0.792)
  BUN | 0.7 (4.15)

39. Primary Outcome: Change From Baseline in pH of Urine at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: The ITT population was used for the analysis. For this particular outcome measure, at week 26, 239 out of 301 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 239
pH | -0.11 (1.065)

40. Primary Outcome: Change From Baseline in Specific Gravity of Urine at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 239
units | 0.0003 (0.00672)

41. Primary Outcome: Change From Baseline in pH of Urine at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: The ITT population was used for the analysis. For this particular outcome measure, at week 52, 195 out of 301 subjects were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 195
pH | -0.09 (1.118)

42. Primary Outcome: Change From Baseline in Specific Gravity of Urine at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 195
units | -0.0010 (0.00695)

43. Primary Outcome: Change From Baseline in Estradiol (E2) Levels at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 243
pg/mL | 0.5 (4.71)

44. Primary Outcome: Change From Baseline in Follicle Stimulating Hormone (FSH) and Luteinizing Hormone (LH) Levels at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 243
IU/L
  FSH | -10.3 (14.13)
  LH | -2.2 (6.86)

45. Primary Outcome: Change From Baseline in Sex Hormone Binding Globulin (SHBG) Levels at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 243
nmol/L | 19.5 (22.67)

46. Primary Outcome: Change From Baseline in Testosterone Levels at Visit 2
Time Frame: Baseline to Week 26 (Visit 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 243
ng/dL
  Testosterone, Free | -0.03 (0.125)
  Testosterone, Total | 1.45 (5.108)

47. Primary Outcome: Change From Baseline in E2 Levels at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 196
pg/mL | 0.4 (10.28)

48. Primary Outcome: Change From Baseline in FSH and LH Levels at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 196
IU/L
  FSH | -15.9 (13.57)
  LH | -1.7 (6.70)

49. Primary Outcome: Change From Baseline in SHBG Levels at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 196
nmol/L | 20.1 (23.19)

50. Primary Outcome: Change From Baseline in Testosterone Levels at Visit 3
Time Frame: Baseline to Week 52 (Visit 3)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Treatment Arm = 60 mg Ospemifene
Number analyzed (Participants) | 196
ng/dL
  Testosterone, Free | 0.00 (0.124)
  Testosterone, Total | 2.23 (5.177)

ADVERSE EVENTS:
Time Frame: 56 weeks
Arm/Group | Treatment Arm = 60 mg Ospemifene
Serious Adverse Events (participants affected / at risk) | 13/301
Other Adverse Events (participants affected / at risk) | 74/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm = 60 mg Ospemifene (N=301)
Acute Myocardial Infarction (Cardiac disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Diverticulitis (Infections and infestations) | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Spinal Meningioma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrahagic Stroke (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety Disorder (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Thrombophlebitis Superficial (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm = 60 mg Ospemifene (N=301)
Sinusitis (Infections and infestations) | 24
Urinary Tract Infection (Infections and infestations) | 26
Hot Flush (Vascular disorders) | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.